CLINICAL TRIAL: NCT07330206
Title: Individualized Treatment Strategies and Long-term Prognosis of Congenital Hydrocephalus: An Integrated Analysis Based on Multicenter Data and Machine Learning
Brief Title: Precision Surgery for Pediatric Hydrocephalus: VPS vs. ETV With ML-Guided Prediction
Acronym: VPS ETV ML
Status: Completed | Type: Observational
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Zhigang Lan, Professor, West China Hospital
Other Study IDs: WestChinaH-HX-2025-011
Record Dates: First submitted 2025-12-29; First posted 2026-01-09 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2024-05

CONDITIONS: Hydrocephalus in Children
Keywords: Ventriculoperitoneal Shunt; Endoscopic Third Ventriculostomy; Machine Learning; Individualized Treatment; Long-term Prognosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ETV group: All undergo endoscopic third ventriculostomy as initial treatment
  Interventions: Diagnostic Test: MRI-Guided Precision Shunt or ETV Strategy
- VPS group: * 320 receive a programmable valve with protocol-driven pressure adjustments
  * 80 receive a fixed-pressure valve (included only in VPS-vs-ETV comparisons, excluded from valve-management sub-analysis)
  Interventions: Diagnostic Test: MRI-Guided Precision Shunt or ETV Strategy

INTERVENTIONS:
Diagnostic Test: MRI-Guided Precision Shunt or ETV Strategy

SUMMARY:
Study type: Multicenter retrospective cohort study with prospective validation Primary purpose: To determine whether an individualized, imaging-guided treatment algorithm Ventriculoperitoneal shunt (VPS) vs endoscopic third ventriculostomy (ETV) improves 2-year neurodevelopmental outcomes in children <18 y with congenital hydrocephalus.

Main questions

* Does ETV produce higher 6-month surgical success and lower 2-year re-intervention rates than VPS in prespecified subgroups (age ≥3 y, obstructive hydrocephalus, normal basal cisterns)?
* Does a machine-learning model (ETV-PS) using pre-operative MRI features accurately predict ETV success (AUC ≥0.80) and thereby reduce unnecessary re-operations?
* Does early, frequent programmable-valve pressure adjustment after VPS decrease over-shunting headaches and improve 2-year cognitive scores compared with standard, infrequent adjustment?

Comparison: ETV group vs. VPS group (1:1 propensity-matched); within VPS cohort, frequent (≥3 adjustments in first 6 mo) vs. infrequent (<3) pressure-tuning arms.

Participants will

* Provide pre-operative clinical data and MRI/CT imaging.
* Undergo either VPS or ETV as clinically indicated; 320 VPS recipients receive programmable valves with protocol-driven pressure logs.
* Return for standardized neurodevelopmental testing Children's Memory Scale (CMS), Wechsler Intelligence Scale for Children(WISC), Pediatric Quality of Life Inventory(PedsQL) and imaging at 6 mo, 1 y and 2 y; valve adjustments tracked electronically.

ELIGIBILITY:
Inclusion Criteria

* Age 0-17.99 years at surgery
* Congenital hydrocephalus confirmed by clinical and MRI/CT findings
* First surgical treatment: either VPS or ETV
* Complete pre-operative MRI/CT and ≥ 2-year follow-up data available

Exclusion Criteria

* Secondary hydrocephalus (tumor, infection, trauma)
* Severe comorbidities affecting neuro-developmental assessment (e.g., major congenital heart disease, genetic-metabolic disorders)
* Incomplete baseline imaging or follow-up < 2 years

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: 800 children ≤17 years with congenital hydrocephalus recruited from 6 tertiary pediatric neurosurgical centers; 1:1 matched VPS (n=400) vs ETV (n=400) cohorts balanced for age, sex, and hydrocephalus subtype.
Sampling Method: Non-Probability Sample
Enrollment: 800 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2024-01-20 (Actual)

PRIMARY OUTCOMES:
Surgical success rate at 6 months post-operation | 6 months
  defined as stable or reduced ventricular volume on MRI/CT without need for re-intervention.

SECONDARY OUTCOMES:
2-year re-intervention rate | 2 years
  any re-operation or shunt revision after
Cognitive improvement | 2 years
  ≥10-point IQ gain or reaching age-appropriate level

CONTACTS AND LOCATIONS:
Locations (1):
- West China Hospital of Sichuan University, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol